CLINICAL TRIAL: NCT03892408
Title: High-flow Nasal Oxygen During Rigid Bronchoscopy Under General Anesthesia: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2019-0005
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2019-03

CONDITIONS: Foreign Bodies; Tumor; Stenosis Trachea; Bronchus Tumour
MeSH Terms: conditions — Foreign Bodies; Neoplasms; Tracheal Stenosis; Bronchial Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective Randomized, open label Trial
Masking Description: triple (Participant, Care Provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optiflow (Experimental): 100 % of oxygen at 70 L / min through Optiflow ™ (Fisher and Paykel Healthcare Limited, Auckland, New Zealand)
  Interventions: Device: Optiflow ™
- Standard (No Intervention): standard anesthesia

INTERVENTIONS:
Device: Optiflow ™ — supply of 100 % of oxygen at 70 L / min through Optiflow ™ (Fisher and Paykel Healthcare Limited, Auckland, New Zealand) plus standard oxygen supply through rigid bronchoscope during apnea period.
  Arms: Optiflow

SUMMARY:
The aim of this study is to evaluate the effect of high-flow nasal cannula oxygen administration on apnea in patients undergoing general anesthesia with rigid bronchoscopy compared with standard anesthesia methods.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing general anesthesia with stent placement or bougination, biopsy or removal of a foreign body or a mass through a rigid bronchoscope
* 2. Patients aged 19 or older who meet American Society of Anesthesiologists (ASA) physical class 2-4

Exclusion Criteria:

* 1. Patients with dementia or cognitive impairment
* 2. pregnant women
* 3. Patients undergoing extracorporeal membrane oxygenation (ECMO)
* 4. Patients with active nasal bleeding), severe nasal obstruction, recent nasal trauma of surgery
* 5. Patients with current maxillofacial trauma or basal skull fracture
* 6. Patients who had previously undergone rigid bronchoscopy / surgery
* 7. If the subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
the lowest oxygen saturation | apnea period during the rigidbroscopic procedure/surgery
  the lowest value of oxygen saturation measured percutaneously at extremity.

SECONDARY OUTCOMES:
Hypoxia occurs the first time | intraoperative (The time taken to reach the point at which peripheral oxygen saturation fell below 90 for the first time immediately after the onset of apnea)
End-tidal carbon dioxide partial pressure | Intraoperative (end-tidal CO2 partial pressure after 3 consecutive breaths after intubation or insertion of laryngeal mask following end of apnea)
Arterial oxygen / carbon dioxide partial pressure | shortly before start of apnea (within 30 seconds)
Arterial oxygen / carbon dioxide partial pressure | shortly after end of apnea (within 30 seconds)
hypoxemia related surgical interruptions | 4) hypoxemia related surgical interruptions during apneic period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine , Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea